CLINICAL TRIAL: NCT01460537
Title: A Phase 1 Study of Copanlisib(Phosphatidylinositol-3 Kinase Inhibitor) in Combination With Gemcitabine (Treatment A) or Cisplatin Plus Gemcitabine (Treatment B) in Subjects With Advanced Solid Malignancy
Brief Title: Phase 1 Study of PI3 (Phosphatidylinositol-3)-Kinase Inhibitor Copanlisib With Gemcitabine or Cisplatin Plus Gemcitabine in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12875
Record Dates: First submitted 2011-09-15; First posted 2011-10-27 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Neoplasms
Keywords: phase I; phosphatidylinositol-3 kinase inhibitor; gemcitabine; cisplatin; maximum tolerated dose
MeSH Terms: conditions — Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A: Gemcitabine-Copanlisib (Experimental): The treatment consists of repetitive cycles, each over 28 days. Treatment continues until disease progression or dose limiting toxicity. If gemcitabine is discontinued for toxicity, Copanlisib may be continued at the discretion of the Investigator if a clinical benefit (response or stable disease for 3 months) is noted. - Hour 0 to 0.5: Gemcitabine (1000 mg/m2 as 30-minute IV infusion) on Days 1, 8 and 15 every 28 days - Hour 1.5 to 2.5: BAY80-6946 (starting dose = 0.6 mg/kg as 60-minute IV infusion, starting 1 hour post completion of gemcitabine infusion) on Days 1, 8 and 15 every 28 days
  Interventions: Drug: Gemcitabine; Drug: BAY80-6946
- Treatment B: Cisplatin-Gemcitabine-Copanlisib (Experimental): Treatment consists of repetitive 21 day cycles for a maximum of 8 cycles. Treatment continues until disease progression, DLT or completion of 8 cycles. After 8 cycles, gemcitabine and Copanlisib, without cisplatin, may continue at the discretion of the Investigator until disease progression or DLT if a clinical benefit is noted (response or stable disease for 3 months). Treatment is administered on Days 1 and 8 every 21 days as follows: - Hour 0 to 1: Cisplatin IV infusion over 60 min (One liter of 0.9% NaCl including 25 mg/m2 cisplatin, 20 mmol of potassium chloride, and 8 mmol of magnesium sulfate) - Hour 1 to 1.5: IV infusion of 500 ml of 0.9% NaCl over 30 min - Hour 1.5 to 2: Gemcitabine (1000 mg/m2 as 30 min IV infusion) - Hour 3 to 4: Copanlisib IV infusion at the MTD determined in Treatment A over 60 min. [If Treatment A MTD is not tolerable, further subject enrollment will begin at one Copanlisib Dose Level lower with the cisplatin-gemcitabine doses remaining constant.]
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: NaCl; Drug: BAY80-6964 fixed dose

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000mg/m2 as 30-minutes IV infusion
Drug: BAY80-6946 — Escalated dose starting from 0.6 mg/kg in 100 mL of 0.9% NaCl as 60-minutes IV infusion
  Arms: Treatment A: Gemcitabine-Copanlisib
Drug: Cisplatin — 1 liter of 0.9% NaCl including 25 mg/m2 cisplatin, 20 mmol of potassium chloride, and 8 nmol of magnesium sulfate over 60 minutes
  Arms: Treatment B: Cisplatin-Gemcitabine-Copanlisib
Drug: NaCl — Infusion of 500 ml of 0.9% NaCl over 30-minutes
  Arms: Treatment B: Cisplatin-Gemcitabine-Copanlisib
Drug: BAY80-6964 fixed dose — BAY80-6946 IV infusion at the maximum tolerated dose determined in Treatment A over 60 min. [If Treatment A MTD is not tolerable, further subject enrollment will begin at one BAY80-6946 Dose Level lower with the cisplatin-gemcitabine doses remaining constant.]
  Arms: Treatment B: Cisplatin-Gemcitabine-Copanlisib

SUMMARY:
This open label Phase I study involves treating subjects with advanced cancer with Copanlisib in combination with either gemcitabine or cisplatin plus gemcitabine. It will determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of Copanlisib in combination with gemcitabine and Copanlisib in combination with cisplatin and gemcitabine. The trial will involve multiple participating sites from the US. Up to a maximum of 70 subjects will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, at least 18 years of age, with advanced or refractory solid tumors in whom gemcitabine (Treatment A) or cisplatin plus gemcitabine (Treatment B) is appropriate medical therapy as determined by the treating physician
* Histological or cytological documentation of non-hematologic, malignant solid tumor, excluding primary brain or spinal tumors, with no current involvement in the CNS
* At least one measurable lesion or evaluable disease, as per RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status Assessment of 0 or 1
* Life expectancy of at least 12 weeks
* Alanine aminotransferase (ALT) ≤ 3.0 x upper limit of normal (ULN; ≤5 x ULN for subjects with liver involvement with cancer)
* Aspartate aminotransferase (AST) ≤ 3.0 x ULN (≤ 5 x ULN for subjects with liver involvement with cancer)
* Total bilirubin ≤ 2.0 x ULN
* Serum creatinine ≤ 1.5 x ULN
* Prothrombin time-international normalized ratio/partial thromboplastin time (PT-INR/PTT) < 1.5 x ULN (Subjects who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists). Low-dose aspirin is permitted (≤ 100 mg daily).

Exclusion Criteria:

* History of cardiac disease congestive; congestive heart failure > New York Heart Association functional classification system (NYHA) Class II; active coronary artery disease, myocardial infarction within 6 months prior to study entry; new onset angina within 3 months prior to study entry or unstable angina, or ventricular cardiac arrhythmias requiring anti-arrhythmic therapy
* Current diagnosis of Type 1 or 2 diabetes mellitus, hyperglycemia (defined as consistent fasting blood glucose > 125 mg/dL) or HgBA1c ≥ 7%
* Use of systemic corticosteroids within 2 weeks of the start of study treatment (topical or inhaled steroids are permitted). Single doses of systemic corticosteroids given as premedication for procedures or non-study drugs may be administered up to 24 hours of first dosing of Copanlisib.
* Poorly controlled hypertension, defined as systolic blood pressure (BP) > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management
* Poorly controlled seizure disorder
* Subjects undergoing renal dialysis
* Use of strong inhibitors of CYP3A4 (eg, ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir, nefazodone and saquinavir) and strong inducers of CYP3A4 (eg, rifampin) are not permitted from Day -14 of Cycle 1 and for the duration of the study.
* Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of first study treatment
* Hormonal therapy during the study or within 2 weeks of first study treatment.
* Bisphosphonate therapy during the first 2 cycles of treatment
* Biological response modifiers, such as granulocyte colony stimulating factor (G-CSF) within 4 weeks of first study treatment
* Radiotherapy to target lesions during study or within 4 weeks of first study treatment
* Known hypersensitivity to the study drugs or active substances or excipients of the preparations
* Use of St John's Wort is prohibited from Day -14 and for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11-18 (Actual); Primary Completion 2015-07-20 (Actual); Study Completion 2015-12-18 (Actual)

PRIMARY OUTCOMES:
Adverse event collection | Up to 3 years or longer if indicated
Maximum tolerated dose, measured by adverse event profile | Up to 3 years or longer if indicated

SECONDARY OUTCOMES:
Maximum drug concentration in plasma (Cmax) of Copanlisib with gemcitabine or cisplatin plus gemcitabine | Approximately 18 months
The time of the maximum concentration (Tmax) of Copanlisib with gemcitabine or cisplatin plus gemcitabine | Approximately 18 months
Area under the curve (AUC) of Copanlisib with gemcitabine or cisplatin plus gemcitabine | Approximately 18 months
Area under the concentration time curve (AUC (0-tn)) of Copanlisib with gemcitabine or cisplatin plus gemcitabine | Approximately 18 months
Half life (t1/2) of Copanlisib with gemcitabine or cisplatin plus gemcitabine | Approximately 18 months
Biomarker evaluation including analysis of pathway activation in tumor tissue and blood/plasma | Up to 3 years or longer if indicated
Tumor Response as measured by RECIST 1.1 criteria | Up to 3 years or longer if indicated

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- United States (3):
  - Tampa, Florida
  - Rochester, Minnesota
  - Chapel Hill, North Carolina